CLINICAL TRIAL: NCT07306520
Title: Effects of the Health Promotion Program on Health Literacy, Physical and Mental Health Status, and Quality of Life of Community Residents in Selected Districts of Gandaki Province, Nepal
Brief Title: Effects of the Health Promotion Program on Health Literacy, Physical and Mental Health Status, and Quality of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, EUN JIN LEE, Professor, Inha University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 241015-1A
Record Dates: First submitted 2025-11-21; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Health Promotion
Keywords: physical health; mental health; chronic disease; quality of life; health literacy; health behavior; health education program; exercise; auricular acupressure; Cohort; health promotion program; Quasi-experimental study; Nepal
MeSH Terms: conditions — Psychological Well-Being; Chronic Disease; Health Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: PRECEDE-PROCEED Model
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Health Education Group (Experimental): Obesity, DM, hypertension, cholesterol
  Interventions: Behavioral: Health education
- Health Education Control Group (No Intervention): Obesity, DM, hypertension, cholesterol
- Auricular Acupressure Group1 (Experimental): Back pain
  Interventions: Device: Auricular acupressure
- Auricular Acupressure Control Group1 (No Intervention): Back pain
- Auricular Acupressure Group2 (Experimental): Dysmenorrhea
  Interventions: Device: Auricular acupressure
- Auricular Acupressure Control Group2 (No Intervention): Dysmenorrhea
- Auricular Acupressure Group3 (Experimental): Perimenopausal symptoms
  Interventions: Device: Auricular acupressure
- Auricular Acupressure Control Group3 (No Intervention): Perimenopausal symptoms
- Exercise Group (Experimental): Obesity, DM, hypertension, cholesterol
  Interventions: Behavioral: Exercise
- Exercise Control Group (No Intervention): Obesity, DM, hypertension, cholesterol

INTERVENTIONS:
Behavioral: Health education — Frequency: 12 sessions, once per week, one hour Will repeat three times a year.
  Arms: Health Education Group
Device: Auricular acupressure — Frequency: 2 sessions, once per week for 2 weeks
  Arms: Auricular Acupressure Group1; Auricular Acupressure Group2; Auricular Acupressure Group3
Behavioral: Exercise — Frequency: 8 sessions, once per week, one hour Will repeat three times a year
  Arms: Exercise Group

SUMMARY:
This study aims to evaluate the physical and mental health status, prevalence of chronic diseases, health literacy, and health behaviors of residents in Gandaki Province, Nepal, and to assess the effectiveness of a community-based health promotion program integrating health education, exercise, and auricular acupressure. The intervention is designed to improve quality of life, health literacy, and chronic disease management among rural populations with limited healthcare access.

This is a prospective interventional cohort study conducted over seven years (2025-2031) in two rural villages of Pokhara, Gandaki Province: Belchautara (experimental) and Rupakot (control). A total of 400 residents aged 19 years and older will be screened and enrolled (200 per village). Participants will be recruited through local nursing colleges and health centers.

Year 1 involves mixed methods research (descriptive-correlational and qualitative) to identify community health needs.

Years 2-7 will employ a quasi-experimental design with annual interventions and follow-up evaluations.

Interventions

1. Health Education Program:

   Frequency: 12 weekly sessions (1 hour each), repeated three times per year. Content: hygiene, nutrition, stress management, lifestyle modification. Measures: health literacy, blood pressure, glucose, cholesterol, anthropometry, quality of life, and PHQ-9.
2. Exercise Program:

   Frequency: 8 weekly sessions (1 hour each), repeated three times per year. Activities: muscle stretching, sit-ups, push-ups, sit-to-stand, and grip strength training.

   Measures: Sit and Reach Test, push-up and sit-up counts, grip strength.
3. Auricular Acupressure:

Indications: back pain, dysmenorrhea, or perimenopausal symptoms. Frequency: once per week for 2 weeks. Measures: Numeric Rating Scale (NRS), Oswestry Disability Index, Menstrual Distress Questionnaire, and Perimenopause Symptom Scale.

Exclusion: pregnancy, metal allergy, or ear disease.

Data will be collected at baseline and post-intervention through structured questionnaires and physical measurements.

ELIGIBILITY:
[Health Screen]:

Inclusion Criteria:

people who

* aged 19 and older
* are able to read and respond to the questionnaire

Exclusion Criteria:

people who are not able to read and respond to the questionnaire

[Health Education]

Inclusion Criteria:

people who

* aged 19 and older
* who are able to read and respond to the questionnaire

Exclusion Criteria:

people who are not able to read and respond to the questionnaire

[Auricular Acupressure]

Inclusion Criteria:

adults ls who reported a pain score of 3 or higher on the Numeric Rating Scale for symptoms (NRS) will be asked about their willingness to participate.

Exclusion Criteria:

* those who are pregnant
* those with a metal allergy
* those with ear-related disorders.

[Exercise]

Inclusion Criteria:

Residents aged 19 and older who are able to read and respond to the questionnaire will be recruited for health screenings and surveys.

Exclusion criteria: Individuals with medical conditions that contraindicate participation in exercise

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-12-25 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Health Literacy (HLS-EU-Q47) | baseline, 12 weeks
  Health literacy will be assessed using the HLS-EU-Q47 (European Health Literacy Survey) developed by the World Health Organization (WHO) European Office. The tool will be used with permission after being translated and adapted by Chun Hee-Ran and Lee Ju-Yeol. It consists of 16 items, including 7 on healthcare, 5 on disease prevention, and 4 on health promotion, measured on a 4-point scale (very difficult to very easy). Responses of difficult/very difficult are scored as 0, while easy/very easy are scored as 1. Higher scores indicate greater health literacy (range 1-16). Based on total scores, 0-8 points indicate inadequate, 9-12 points indicate borderline, and 13 points or higher indicate sufficient health lieteracy.
Subjective Perception of Health (5-point Likert scale) | baseline, 12 weeks
  Subjective perception of health refers to an individual's self-assessment of their health status, whether good or poor. This is evaluated on a 5-point Likert scale with the responses: ① Very good, ② Good, ③ Fair, ④ Poor, and ⑤ Very poor. The subjective change in health status is a self-assessment of whether one's health has improved or worsened compared to a previous assessment. The question is: "How is your current health compared to the previous baseline survey?" Responses are measured on a 5-point Likert scale: ① Very much improved, ② Somewhat improved, ③ Same as before, ④ Somewhat worsened, and ⑤ Very much worsened (16).
Mental Health (Patient Health Questionnaire (PHQ-9)) | baseline, 12 weeks
  The PHQ-9 (Patient Health Questionnaire) will assess the Mental Health. The PHQ-9 is a tool developed for diagnosing major depressive disorder and is widely used in primary healthcare settings. Participants are asked how often they experienced problems over the past two weeks, measured on a 4-point scale (Not at all to Nearly every day), with scores ranging from 0-27. Higher scores indicate more severe depressive symptoms. When using a cutoff score of 10, the sensitivity (94%) and specificity (80%) are high. Cronbach's alpha was reported as 0.84 among 125 Nepali primary care patients.
Quality of life (EQ-5D-5L Score) | baseline, 12 weeks
  Quality of life will be measured using the EQ-5D-5L, developed and translated in Nepalese by EuroQol. The EQ-5D-5L assesses current health status across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a 5-point scale from no problems to extreme problems. Reliability (ICC = 0.75). and one factor explained 88.3% of total variance. The EuroQol group provides a Nepali version of the tool, which will be used with approval.

SECONDARY OUTCOMES:
Numeric Rating Scale for Symptoms (NRS) | baseline, 12 weeks
  The Numeric Rating Scale for symptoms (NRS) is widely used in clinical practice due to its simplicity and convenience for assessing pain and various symptoms. The NRS measures symptoms on a scale from 0 to 10, with scores closer to 10 indicating greater severity of perceived symptoms.
Blood Pressure (automatic blood pressure cuff) | baseline, 12 weeks
  Blood pressure will be measured using an automatic blood pressure cuff. Both systolic and diastolic blood pressure will be measured. Participants will be asked to sit quietly for 2-3 minutes and remove any tight clothing. Measurements will be taken on both the right and left arms, ensuring that the mid-arm is positioned at heart level. Elevated blood pressure is defined as exceeding the 95th percentile for age and height.
Fasting blood glucose level | baseline, 12 weeks
  To measure fasting capillary blood glucose, participants will be instructed to fast overnight after dinner. The next morning, their fingers will be disinfected with alcohol swabs, allowed to dry, and blood will be drawn from peripheral capillaries using a new lancet. Measurements will be taken using the Accu-Chek Active glucose meter and the SD CodeFree glucose meter.
Fasting Cholesterol Level | baseline, 12 weeks
  To measure fasting cholesterol, participants will be instructed to fast overnight after dinner. The next morning, their fingers will be disinfected with alcohol swabs, allowed to dry, and blood will be drawn from peripheral capillaries using a new lancet. Measurements will be taken using the CardioCheck PA device.
Effect of exercise (SIt-and-Reach Test Score) | baseline, 8 weeks
  The Sit-and-Reach Test will be used for the effect of exercise. This test is a simple, widely used method to assess overall flexibility, particularly of the lower back and hamstrings. It involves reaching forward while seated with legs straight, measuring the distance reached. Participants sit on the floor with their legs fully extended and feet placed against a standardized measurement box. With both hands overlapped and arms fully extended, participants reach forward as far as possible and hold the position for 2 seconds. The distance reached (in centimeters) is recorded as the Sit-and-Reach Test score, with higher values indicating greater flexibility.
Effect of exercise (Grip Strength Test) | baseline, 8 weeks
  This test will be used for the effect of exercise. Grip strength test measures how much force a person can exert when squeezing a hand grip dynamometer. It's a simple and commonly used method for assessing general muscle strength, particularly in the forearm, and is often used in medical and fitness settings. Grip strength is measured using an electronic hand dynamometer. Participants hold the dynamometer in their both hands separately, with the arm in a neutral position alongside the body. They are instructed to squeeze the device with maximum effort for a few seconds. The highest value (in kilograms) from repeated trials is recorded as the final grip strength score.
Effect of exercise (Push-up and Sit-up Test (1-Minute Test)) | baseline, 8 weeks
  This test will be used for the effect of exercise. Muscular endurance is assessed by counting the number of push-ups and sit-ups performed within one minute. For push-ups, participants perform standard push-ups with proper posture. For sit-ups, participants lie in the supine position with knees bent and perform consecutive sit-ups for one minute. The total number of correctly completed repetitions within 60 seconds is recorded for each exercise.
Dysmenorrhea (Menstrual Distress Questionnaire (MEDI-Q)) | baseline, 2 weeks
  Dysmenorrhea will be measured using the Menstrual Distress Questionnaire (MEDI-Q). This tool developed by Silvia et al. 2021 assess 25 items, covering the following areas: pain, discomfort, psychic or cognitive changes, gastrointestinal symptoms and changes in physiological functions. The MEDI-Q Total Score is obtained from the sum of all the distress scores calculated for each item. The minimum score obtainable is 0, indicating the absence of any specified symptom relevant to generate distress during menstruation in the previous 12 months. The maximum score is 125, indicating the presence of all the investigated symptoms in more than one-half of menstruations in the past year, each of them generating severe distress. This tool has high internal consistency (Cronbach's alpha ≥0.95) and test-retest reliability (from 0.60 to 0.70).
Perimenopause symptoms (Perimenopausal Symptoms Rating Scale (MRS scale)) | baseline, 2 weeks
  Perimenopause symptoms will be measured using the Perimenopausal Symptoms Rating Scale. This tool will be used in this study which is a valuable tool for assessing health related quality of life of women in the menopausal transition and it is used worldwide. It is a standardized scale meeting psychometric norm. There are 11 questions and each symptom has five ordinal scales of rating menopausal symptoms by its severity. Severity is described into five levels as none (0), mild (1), moderate (2), severe (3) and very severe (4). For this study, the tool will be used with permission and applied in its validated Nepali version, which has been previously used in Nepal (Menopause Rating Scale: Validation and Applicability in Nepalese Women).
Disability in daily life due to musculoskeletal pain (Oswestry Disability Index(ODI)) | baseline. 2 weeks
  The level of disability in daily life due to musculoskeletal pain was measured using the Oswestry Disability Index. The ODI consists of 10 Items (pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual activity, social life, and traveling), with each item scored from 0 to 5. The total score is summed and then multiplied by 2 to convert it into a percentage. The levels of disability are interpreted as follows - 0-20%: Minimal disability (able to perform daily activities without special measures), 21-40%: Moderate disability (pain and difficulty present in daily life, requiring conservative treatment), 41-60%: Severe disability (persistent pain significantly interferes with daily life, requiring detailed examination), 61-80%: Crippling disability (affects all aspects of personal life, requiring active treatment), 81-100%: Bed-bound (unable to carry out daily activities)

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea